CLINICAL TRIAL: NCT02923453
Title: Efficacy and Safety of American Ginseng (Penax Quinquefolius) Extract on Glycemic Control in Individuals With Type 2 Diabetes: A Double-blind, Randomized, Crossover Clinical Trial
Brief Title: Effect of Ginseng in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNT 2000
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Type II Diabetes Control

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1g/meal of placebo three times per day (3g/day) for 8-weeks.
  Interventions: Dietary Supplement: Placebo
- Ginseng Extract (Active Comparator): CNT2000 (Chai-Na- Ta Corp., Langley, BC) American ginseng extract 1g/meal of placebo three times per day (3g/day) for 8-weeks.
  Interventions: Dietary Supplement: CNT 2000 American ginseng extract

INTERVENTIONS:
Dietary Supplement: CNT 2000 American ginseng extract
  Arms: Ginseng Extract
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Objective: We aim to evaluate longer term efficacy and safety of AG as an add-on therapy in patients with type 2 diabetes controlled by conventional treatment. Materials and Methods: A total of 23 type 2 patients are enrolled in the study. Utilizing a double-blind, crossover design, the participants are randomized to receive either placebo or American ginseng extract (AG) 1g/meal=3g/day for 8-week, while maintained on their conventional diabetes treatment. Following ≥4-week washout period the participants are crossed over to another 8-week treatment arm. Throughout the study period, all individuals maintain their original diabetes treatment and regular lifestyle. The primary endpoint is HbA1c, and secondary are fasting blood glucose and insulin, blood pressure, serum nitrates/nitrites (NOx) and PAI-1. Safety parameters include liver, kidney and hemostatic functions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of type 2 diabetes of ≥1 year duration
* BMI between 25-35kg/m^2
* HbA1c between 6.5-8.5%

Exclusion Criteria:

* Patients on insulin therapy
* Impaired hepatic or renal function
* Clinically manifested diabetic complications
* Present cardiac problems
* Uncontrolled hypoglycemia
* Cigarette smokers
* Alcohol consumption (>2 drinks per week)
* Taking ginseng or other herb with possible hypoglycemic effect
* Involvement in any other investigational drug studies
* Changed medication during the course of the study periods or during the washout period

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1998-03; Primary Completion 2001-12 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 8 weeks

SECONDARY OUTCOMES:
Fasting blood glucose | 8 weeks
Fasting blood insulin | 8 weeks
Blood pressure | 8 weeks
serum nitrates/nitrites (NOx) | 8 weeks
Plasminogen activator inhibitor-1 (PAI-1) | 8 weeks
Alanine amino-transferase (ALT) | 8 weeks
serum creatinine | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- : Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Van Gaal L, Scheen A. Weight management in type 2 diabetes: current and emerging approaches to treatment. Diabetes Care. 2015 Jun;38(6):1161-72. doi: 10.2337/dc14-1630. PMID 25998297
- [Background] Bacon L, Aphramor L. Weight science: evaluating the evidence for a paradigm shift. Nutr J. 2011 Jan 24;10:9. doi: 10.1186/1475-2891-10-9. PMID 21261939
- [Background] Bravata DM, Sanders L, Huang J, Krumholz HM, Olkin I, Gardner CD, Bravata DM. Efficacy and safety of low-carbohydrate diets: a systematic review. JAMA. 2003 Apr 9;289(14):1837-50. doi: 10.1001/jama.289.14.1837. PMID 12684364
- [Background] Dansinger ML, Gleason JA, Griffith JL, Selker HP, Schaefer EJ. Comparison of the Atkins, Ornish, Weight Watchers, and Zone diets for weight loss and heart disease risk reduction: a randomized trial. JAMA. 2005 Jan 5;293(1):43-53. doi: 10.1001/jama.293.1.43. PMID 15632335
- [Background] Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, McManus K, Champagne CM, Bishop LM, Laranjo N, Leboff MS, Rood JC, de Jonge L, Greenway FL, Loria CM, Obarzanek E, Williamson DA. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009 Feb 26;360(9):859-73. doi: 10.1056/NEJMoa0804748. PMID 19246357
- [Background] Post RE, Mainous AG 3rd, King DE, Simpson KN. Dietary fiber for the treatment of type 2 diabetes mellitus: a meta-analysis. J Am Board Fam Med. 2012 Jan-Feb;25(1):16-23. doi: 10.3122/jabfm.2012.01.110148. PMID 22218620
- [Background] Johnston BC, Kanters S, Bandayrel K, Wu P, Naji F, Siemieniuk RA, Ball GD, Busse JW, Thorlund K, Guyatt G, Jansen JP, Mills EJ. Comparison of weight loss among named diet programs in overweight and obese adults: a meta-analysis. JAMA. 2014 Sep 3;312(9):923-33. doi: 10.1001/jama.2014.10397. PMID 25182101
- [Background] Buckley JD, Howe PRC. Long-chain omega-3 polyunsaturated fatty acids may be beneficial for reducing obesity-a review. Nutrients. 2010 Dec;2(12):1212-1230. doi: 10.3390/nu2121212. Epub 2010 Dec 9. PMID 22254005
- [Background] Valdivia-Lopez MA, Tecante A. Chia (Salvia hispanica): A Review of Native Mexican Seed and its Nutritional and Functional Properties. Adv Food Nutr Res. 2015;75:53-75. doi: 10.1016/bs.afnr.2015.06.002. Epub 2015 Aug 5. PMID 26319904
- [Background] Vuksan V, Whitham D, Sievenpiper JL, Jenkins AL, Rogovik AL, Bazinet RP, Vidgen E, Hanna A. Supplementation of conventional therapy with the novel grain Salba (Salvia hispanica L.) improves major and emerging cardiovascular risk factors in type 2 diabetes: results of a randomized controlled trial. Diabetes Care. 2007 Nov;30(11):2804-10. doi: 10.2337/dc07-1144. Epub 2007 Aug 8. PMID 17686832
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Bazinet RP, McMillan EG, Cunnane SC. Dietary alpha-linolenic acid increases the n-3 PUFA content of sow's milk and the tissues of the suckling piglet. Lipids. 2003 Oct;38(10):1045-9. doi: 10.1007/s11745-006-1159-9. PMID 14669969
- [Background] Katsuki A, Urakawa H, Gabazza EC, Murashima S, Nakatani K, Togashi K, Yano Y, Adachi Y, Sumida Y. Circulating levels of active ghrelin is associated with abdominal adiposity, hyperinsulinemia and insulin resistance in patients with type 2 diabetes mellitus. Eur J Endocrinol. 2004 Nov;151(5):573-7. doi: 10.1530/eje.0.1510573. PMID 15538935
- [Background] Chandran M, Phillips SA, Ciaraldi T, Henry RR. Adiponectin: more than just another fat cell hormone? Diabetes Care. 2003 Aug;26(8):2442-50. doi: 10.2337/diacare.26.8.2442. No abstract available. PMID 12882876
- [Background] Guo Y, Ma L, Enriori PJ, Koska J, Franks PW, Brookshire T, Cowley MA, Salbe AD, Delparigi A, Tataranni PA. Physiological evidence for the involvement of peptide YY in the regulation of energy homeostasis in humans. Obesity (Silver Spring). 2006 Sep;14(9):1562-70. doi: 10.1038/oby.2006.180. PMID 17030967
- [Background] Stenlof K, Rossner S, Vercruysse F, Kumar A, Fitchet M, Sjostrom L; OBDM-003 Study Group. Topiramate in the treatment of obese subjects with drug-naive type 2 diabetes. Diabetes Obes Metab. 2007 May;9(3):360-8. doi: 10.1111/j.1463-1326.2006.00618.x. PMID 17391164
- [Background] Hensrud DD. Dietary treatment and long-term weight loss and maintenance in type 2 diabetes. Obes Res. 2001 Nov;9 Suppl 4:348S-353S. doi: 10.1038/oby.2001.141. PMID 11707564
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycemia in type 2 diabetes, 2015: a patient-centered approach: update to a position statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2015 Jan;38(1):140-9. doi: 10.2337/dc14-2441. No abstract available. PMID 25538310
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Vilsboll T, Zdravkovic M, Le-Thi T, Krarup T, Schmitz O, Courreges JP, Verhoeven R, Buganova I, Madsbad S. Liraglutide, a long-acting human glucagon-like peptide-1 analog, given as monotherapy significantly improves glycemic control and lowers body weight without risk of hypoglycemia in patients with type 2 diabetes. Diabetes Care. 2007 Jun;30(6):1608-10. doi: 10.2337/dc06-2593. Epub 2007 Mar 19. No abstract available. PMID 17372153
- [Background] Nieman DC, Cayea EJ, Austin MD, Henson DA, McAnulty SR, Jin F. Chia seed does not promote weight loss or alter disease risk factors in overweight adults. Nutr Res. 2009 Jun;29(6):414-8. doi: 10.1016/j.nutres.2009.05.011. PMID 19628108
- [Background] Ayerza R, Coates W. Dietary levels of chia: influence on yolk cholesterol, lipid content and fatty acid composition for two strains of hens. Poult Sci. 2000 May;79(5):724-39. doi: 10.1093/ps/79.5.724. PMID 10824962
- [Background] Ayerza R. The seed's protein and oil content, fatty acid composition, and growing cycle length of a single genotype of chia (Salvia hispanica L.) as affected by environmental factors. J Oleo Sci. 2009;58(7):347-54. doi: 10.5650/jos.58.347. PMID 19491529
- [Background] Vuksan V, Jenkins AL, Dias AG, Lee AS, Jovanovski E, Rogovik AL, Hanna A. Reduction in postprandial glucose excursion and prolongation of satiety: possible explanation of the long-term effects of whole grain Salba (Salvia Hispanica L.). Eur J Clin Nutr. 2010 Apr;64(4):436-8. doi: 10.1038/ejcn.2009.159. Epub 2010 Jan 20. PMID 20087375
- [Background] Nieman DC, Gillitt N, Jin F, Henson DA, Kennerly K, Shanely RA, Ore B, Su M, Schwartz S. Chia seed supplementation and disease risk factors in overweight women: a metabolomics investigation. J Altern Complement Med. 2012 Jul;18(7):700-8. doi: 10.1089/acm.2011.0443. PMID 22830971
- [Background] Sahakyan KR, Somers VK, Rodriguez-Escudero JP, Hodge DO, Carter RE, Sochor O, Coutinho T, Jensen MD, Roger VL, Singh P, Lopez-Jimenez F. Normal-Weight Central Obesity: Implications for Total and Cardiovascular Mortality. Ann Intern Med. 2015 Dec 1;163(11):827-35. doi: 10.7326/M14-2525. Epub 2015 Nov 10. PMID 26551006
- [Background] Rao AD, Milbrandt EB. To JUPITER and beyond: statins, inflammation, and primary prevention. Crit Care. 2010;14(3):310. doi: 10.1186/cc9006. Epub 2010 May 13. No abstract available. PMID 20497597
- [Background] Kinlay S. Low-density lipoprotein-dependent and -independent effects of cholesterol-lowering therapies on C-reactive protein: a meta-analysis. J Am Coll Cardiol. 2007 May 22;49(20):2003-9. doi: 10.1016/j.jacc.2007.01.083. Epub 2007 May 4. PMID 17512355
- [Background] Ridker PM, Rifai N, Rose L, Buring JE, Cook NR. Comparison of C-reactive protein and low-density lipoprotein cholesterol levels in the prediction of first cardiovascular events. N Engl J Med. 2002 Nov 14;347(20):1557-65. doi: 10.1056/NEJMoa021993. PMID 12432042
- [Background] Jenkins DJ, Kendall CW, Vuksan V. Viscous fibers, health claims, and strategies to reduce cardiovascular disease risk. Am J Clin Nutr. 2000 Feb;71(2):401-2. doi: 10.1093/ajcn/71.2.401. No abstract available. PMID 10648250
- [Background] Roberfroid MB. Inulin-type fructans: functional food ingredients. J Nutr. 2007 Nov;137(11 Suppl):2493S-2502S. doi: 10.1093/jn/137.11.2493S. PMID 17951492
- [Background] Detopoulou P, Panagiotakos DB, Chrysohoou C, Fragopoulou E, Nomikos T, Antonopoulou S, Pitsavos C, Stefanadis C. Dietary antioxidant capacity and concentration of adiponectin in apparently healthy adults: the ATTICA study. Eur J Clin Nutr. 2010 Feb;64(2):161-8. doi: 10.1038/ejcn.2009.130. Epub 2009 Nov 11. PMID 19904292
- [Background] Mohammadi E, Rafraf M, Farzadi L, Asghari-Jafarabadi M, Sabour S. Effects of omega-3 fatty acids supplementation on serum adiponectin levels and some metabolic risk factors in women with polycystic ovary syndrome. Asia Pac J Clin Nutr. 2012;21(4):511-8. PMID 23017309
- [Background] Vuksan V, Rogovik AL, Jovanovski E, Jenkins AL. Fiber facts: benefits and recommendations for individuals with type 2 diabetes. Curr Diab Rep. 2009 Oct;9(5):405-11. doi: 10.1007/s11892-009-0062-1. PMID 19793511
- [Background] Wanders AJ, van den Borne JJ, de Graaf C, Hulshof T, Jonathan MC, Kristensen M, Mars M, Schols HA, Feskens EJ. Effects of dietary fibre on subjective appetite, energy intake and body weight: a systematic review of randomized controlled trials. Obes Rev. 2011 Sep;12(9):724-39. doi: 10.1111/j.1467-789X.2011.00895.x. Epub 2011 Jun 16. PMID 21676152
- [Background] Jiao J, Xu JY, Zhang W, Han S, Qin LQ. Effect of dietary fiber on circulating C-reactive protein in overweight and obese adults: a meta-analysis of randomized controlled trials. Int J Food Sci Nutr. 2015 Feb;66(1):114-9. doi: 10.3109/09637486.2014.959898. Epub 2015 Jan 12. PMID 25578759
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Derived] Vuksan V, Xu ZZ, Jovanovski E, Jenkins AL, Beljan-Zdravkovic U, Sievenpiper JL, Mark Stavro P, Zurbau A, Duvnjak L, Li MZC. Efficacy and safety of American ginseng (Panax quinquefolius L.) extract on glycemic control and cardiovascular risk factors in individuals with type 2 diabetes: a double-blind, randomized, cross-over clinical trial. Eur J Nutr. 2019 Apr;58(3):1237-1245. doi: 10.1007/s00394-018-1642-0. Epub 2018 Feb 24. PMID 29478187